CLINICAL TRIAL: NCT04134351
Title: Does Sphingosine-1-phosphate Constrict Human Airways? In-vivo Challenge Pilot Study.
Brief Title: Sphingosine-1-phosphate in Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 223069
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Bronchial challenge test — Bronchial challenge test with sphingosine-1-phosphate

SUMMARY:
This study is being undertaken in order to enhance our understanding how human airways are being constricted in healthy people and in individuals with asthma. There is an unmet need for identification of new pathways (mediators) related to enhanced constriction of the asthmatic airways that would reveal new targets for therapy. Sphingosine-1-phosphate (S1P) is a naturally occurring bioactive lipid molecule that has been suggested to play an important role in asthma. Physiologically, S1P can be detected in human blood but local tissue concentrations (for example in the lung) are very low. Upon activation many cells can secrete S1P. Increased concentrations of S1P have been detected in airways of asthmatic subjects after allergen inhalation. When studied in animal models, S1P did not cause contraction of airways in healthy animals but contracted airways in animal with pulmonary inflammation. In laboratory experiments S1P has been shown to be a potent constrictor of cells responsible for contraction of human airways. As yet, however, we lack evidence that S1P actually causes constriction of airways in real life. Establishing S1P as a molecule capable of causing airway constriction in humans and perhaps specifically in asthmatics will have important implications for our understanding of physiological and pathophysiological responses in human airways and could open new windows for therapeutic strategies in diseases like asthma.

ELIGIBILITY:
Cases (asthmatics) inclusion criteria

1. Physician diagnosed asthma, defined as a clear history of typical symptoms and clear reversibility of the PEF/FEV1 (12% or more) within the past year and/or methacholine PC20 < 8mg/ml.

Cases Exclusion criteria

1. Pregnancy or lactation
2. Moderate / Severe asthma (FEV1/PEF < 80%of the predicted value at screening)
3. Patients with any chronic illness other than asthma and other recognised atopic diseases (eczema, rhinitis) or any other abnormality which in the opinion of the principal investigator might compromise the study findings
4. A history of recent (within the past 4 weeks) upper or lower respiratory tract infection
5. Patients receiving oral, inhaled or parenteral glucocorticoid therapy (steroid) within the last 4 weeks, long acting relievers (salmeterol, formoterol) and antileukotrienes (montelukast) within last 72 hours.
6. Inadequate contraception in women of childbearing age
7. Inability to comprehend or comply with the protocol

Controls inclusion criteria

1. Lifelong absence of asthma symptoms and lung function within the normal range.

Controls exclusion criteria

1. Pregnancy or lactation
2. Patients with any chronic illness or any other abnormality which in the opinion of the principal investigator might compromise the study findings
3. A history of recent (within the past 4 weeks) upper or lower respiratory tract infection
4. Oral, inhaled or parenteral glucocorticoid therapy (steroid) within the last 4 weeks, long acting relievers (salmeterol, formoterol) and antileukotrienes (montelukast) within last 72 hours
5. Inadequate contraception in women of childbearing age
6. Inability to comprehend or comply with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-02-22 (Estimated); Study Completion 2022-02-22 (Estimated)

PRIMARY OUTCOMES:
Bronchoconstriction | 1 hour after challenge
  Bronchoconstriction in response to challenge measured by spirometry (FEV1)(PC20)

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Woszczek, MD, PhD, Principal Investigator — King's College London
Locations (1):
- Allergy Day Care Unite, Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No